CLINICAL TRIAL: NCT00167921
Title: A Multiple-Dose, Comparative Bioavailability Study of Premarin® Vaginal Cream Versus Premarin® Oral Tablets in Postmenopausal Women With Atrophic Vaginitis.
Brief Title: Study Comparing Premarin® Vaginal Cream Versus Premarin® Oral Tablets in Atrophic Vaginitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 0713S5-414
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2007-05-28 (Estimated); Status verified 2007-05

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Premarin® Vaginal Cream
Drug: Premarin® oral tablets

SUMMARY:
The purpose of this study is to characterize the systemic exposure and bioavailability at steady state of Premarin® Vaginal Cream compared with Premarin® oral tablets in postmenopausal women with atrophic vaginitis.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy postmenopausal women.
* Intact uterus.
* Clinical diagnosis of moderate to severe atrophic vaginitis.

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2005-10

PRIMARY OUTCOMES:
To characterize the systemic exposure and bioavailability at steady state of Premarin® Vaginal Cream compared with oral Premarin® tablets in postmenopausal women with atrophic vaginitis.

SECONDARY OUTCOMES:
To estimate the systemic exposure in postmenopausal women taking a typical regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (2):
- United States (2):
  - Miami, Florida
  - Baltimore, Maryland